CLINICAL TRIAL: NCT06282692
Title: An Open Label, Phase III Clinical Trial (Immunobridging Study) of INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated)) in Healthy Population Aged 12 to 17 Years Old
Brief Title: INAVAC Vaccine Phase III (Immunobridging Study) in Healthy Population Aged 12 to 17 Years Old
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Indonesia-MoH (Other Government); Universitas Airlangga (Other); PT Biotis Pharmaceuticals, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNAIR-MP-INAKTIF-R-005
Record Dates: First submitted 2023-06-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pandemic; COVID-19 Vaccines
Keywords: Inactivated COVID-1 9 Vaccine; Immunogenicity; Safety; COVID-19; Indonesia; Immunobridging Study
MeSH Terms: conditions — COVID-19 | interventions — vaksin merah putih - UA SARS-CoV-2 COVID-19 vaccine

STUDY DESIGN:
Masking Description: This is an open label, phase III trial - immunobridging study. There will be only 1 group in the study. All subjects (12 to 17 years old) will receive INAVAC 5 µg dose.
  The vaccine will be administered with 2-dose schedule, intramuscularly, with 28 day interval.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: (Experimental): INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated) 5 µg
  Study product are provided in the form of liquid in vial single dose (0.5 ml). The vaccine will be given 1 dose (0.5 ml) twice.
  Interventions: Biological: INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated) 5 µg

INTERVENTIONS:
Biological: INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated) 5 µg — Dose : 1 dose 0.5 ml containing 5 µg inactivated SARS-CoV-2 virus, Tween 80, histidine, Polysorbate 80, Aluminium hydroxide gel, and sodium chloride.

SUMMARY:
This is an open label, phase III trial - immunobridging study. There will be only 1 group in the study. All subjects (12 to 17 years old) will receive INAVAC 5 µg dose. The vaccine will be administered with 2-dose schedule, intramuscularly, with 28 day interval. All subjects will be followed for 12 months.

INAVAC is an inactivated vaccine made of SARS-CoV-2 virus isolated from a patient in Surabaya, composed with aluminium hydroxy gel, tween 80, and L-histidine, and this study will be the first phase III in adolescents.

DETAILED DESCRIPTION:
This is an open label, phase III trial - immunobridging study. There will be only 1 group in the study. All subjects (12 to 17 years old) will receive INAVAC 5 µg dose. The vaccine will be administered with 2-dose schedule, intramuscularly, with 28 day interval. All subjects will be followed for 12 months.

This study will have three interim and one full analysis The main focus is immunogenicity and safety or reactogenicity issues.

Data Safety Monitoring Board will be commissioned for this study to evaluate safety data over the study period and to review any events that meet a specific study pausing rule or any other safety issue that may arise. They will review the 7 and 28 days safety data following the first dose of vaccine, and then the 7 and 28 days after the second dose. The immunogenicity data will be evaluated until 12 months after the second dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adolescents, age 12 to 17 years old, males and females. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
2. Subjects and the parents or guardians have been informed properly regarding the study and signed the informed consent and assent forms
3. Subject and the parents or guardians will commit to comply with the instructions of the investigator and the schedule of the trial
4. Participants agree not to donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine.
5. Subjects and the parents or guardians must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another vaccine trial
2. Evolving mild, moderate, and severe illness, especially infectious diseases or fever (axillary temperature 37.5oC or more) concurrent or within 7 days prior to first study vaccination. This includes respiratory or constitutional symptms consistent with SARS-CoV-2 (cough, sore throat, difficulty in breathing, etc)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Any autoimmune or immunodeficiency disease/condition
6. Subjects who have received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived products, long term corticosteroid - more than 2 weeks, and so on), OR anticipation of the need for immunosuppressive treatment within 6 months after last vaccination. The use of topical or nasal steroid will be permitted.
7. Unstable chronic disease, inclusive of uncontrolled hypertension, congestive heart failure, chronic obstructive pulmonary disease, asthma, chronic urticaria, diabetes requiring use of medicine. The final decision regarding this condition will be decided by the attending field clinicians or investigator.
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
9. Individuals who previously receive any vaccines against Covid-19
10. Subjects already immunized with any vaccine within 4 weeks prior and expect to receive other vaccines within 60 days following the first dose
11. Individuals who have a previously ascertained Covid-19 in the period of 1 month (for mild, moderate, or asymptomatic people) or 3 months (for severe Covid-19) before the first recruit of this study, or in a close contact in the last 14 days with confirmed case of Covid-19.
12. Positive test for SARS-CoV-2 (Antigen test or, if necessary, PCR test) at screening prior to first vaccination. Testing may be repeated during the screening period if exposure to positive confirmed case of SARS-CoV-2 is suspected, at the discretion of investigator.
13. Alcohol or substance abuse
14. HIV patients.
15. Malignancy patients within 2 years prior to first study vaccination.
16. Any neurological disease or history of significant neurological disorder such as meningitis, encephalitis, Guillain-Barre Syndrome, multiple sclerosis, etc
17. Vital sign abnormalities and clinical laboratory abnormalities as decided by the investigators. Vital sign measurements and clinical laboratory testing may be repeated before the final decision.
18. Women who are pregnant or who plan to become pregnant during the study.
19. Participant has major psychiatric problem or illness
20. Participant cannot communicate reliably with the investigator
21. Participant has contraindication to intramuscular injection and blood draws, such as bleeding disorders or phobia.
22. Participant had major surgery within 12 weeks before vaccination which will not be fully recovered, or has major surgery planned during the time participant is expected to participate in the study or within 6 months after the last dose of study vaccine administration.
23. Any condition that in the opinion of the investigators would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine or interpretation of the study results
24. Study team members.
25. Subject planning to move from the study area before the end of study period.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
Vaccine Neutralizing Antibody Profile | 28 days after two doses vaccination of INAVAC.
  SARS-CoV-2 neutralizing titers in serum measured by a virus neutralization assay, at 28 days after two doses vaccination of INAVAC in healthy adolescents age 12 to 17 years old, compared with previous results in adults with two doses of similar vaccine (phase 3 in adults).

SECONDARY OUTCOMES:
Incidence of Adverse Events | 30 minutes, 24 hours, 7 and 28 days following the first dose and 30 minutes, 24 hours, 7 and 28 days, 3, 6 and 12 months after the second doses of INAVAC
  1. Solicited - clinical (local and systemic) adverse events for 30 minutes, 24 hours, 7 and 28 days after the first and second vaccination, and then 3, 6, and 12 months after the second injection of INAVAC in healthy adolescents age 12 to 17 years old, compared with previous results in adults with two doses of similar vaccine (phase 3 in adults).
  2. Unsolicited adverse events for 30 minutes, 24 hours, 7 and 28 days after the first and second vaccination, and then 3, 6, and 12 months after the second injection of INAVAC in healthy adolescents age 12 to 17 years old, compared with previous results in adults with two doses of similar vaccine (phase 3 in adults).
  3. Serious adverse event (SAE) throughout the study (from the first vaccination).
Humoral Immunogenicity - The Neutralizing Antibody Titers in Serum | 3, 6, and 12 months, following vaccination with two doses of INAVAC
  Evaluate SARS-Cov-2 neutralizing titers in serum measured by virus neutralization assay at 3, 6, and 12 months, following vaccination with two doses of INAVAC in healthy adolescents age 12 to 17 years old, compared with previous results in adults with two doses of similar vaccine (phase 3 in adults).
Humoral Immunogenicity - Levels of SARS-CoV-2 Binding Antibodies by CLIA | 28 days, 3, 6, and 12 months after the second vaccination of INAVAC
  SARS-CoV-2 binding antibodies measured by CLIA: analysis of antibodies binding to the SARS-CoV-2 S-protein.
Cellular Immunogenicity Profile | 28 days, 3, 6, and 12 months, following vaccination with two doses of INAVAC
  1. Th1 immune responses assessed by Flow cytometri
  2. Th2 immune responses assessed by Flow cytometri
Persistence of Antibody Level | 12 months after the second injection
  Evaluate the persistence of antibody level over time for 12 months after second injection.
Whole Genome Sequencing (WGS) of SARS-CoV-2 | Throughout the study, an average of 1 year
  Whole genome sequencing (WGS) of S protein of SARS-CoV-2 virus from all positive Covid-19 cases

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, MD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Wang Z, Wang G, Lau JY, Zhang K, Li W. COVID-19 in early 2021: current status and looking forward. Signal Transduct Target Ther. 2021 Mar 8;6(1):114. doi: 10.1038/s41392-021-00527-1. PMID 33686059
- [Background] Noh JY, Song JY, Yoon JG, Seong H, Cheong HJ, Kim WJ. Safe hospital preparedness in the era of COVID-19: The Swiss cheese model. Int J Infect Dis. 2020 Sep;98:294-296. doi: 10.1016/j.ijid.2020.06.094. Epub 2020 Jun 30. PMID 32619759
- [Background] New York Vaccine Tracker. Downloaded from https://www.nytimes.com/interactive/2020/science/coronavirus-vaccinetracker.html. Accessed 11 April 2022.
- [Background] Badan POM Republik Indonesia. Dowloaded from https://www.pom.go.id/new/view/more/pers/605/Pastikan-Keamanan-danMutu-Vaksin---Badan-POM-Kawal-Uji-Klinik-Vaksin-Merah-Putih.html. Accessed 11 October 2021.
- [Background] Irwin A. What it will take to vaccinate the world against COVID-19. Nature. 2021 Apr;592(7853):176-178. doi: 10.1038/d41586-021-00727-3. No abstract available. PMID 33767468
- [Background] So AD, Woo J. Reserving coronavirus disease 2019 vaccines for global access: cross sectional analysis. BMJ. 2020 Dec 15;371:m4750. doi: 10.1136/bmj.m4750. PMID 33323376
- [Background] Worldometer coronavirus cases. Downloaded from https://www.worldometers.info/coronavirus/. Accessed 11 October 2021.
- [Background] Biswas M, Rahaman S, Biswas TK, Haque Z, Ibrahim B. Association of Sex, Age, and Comorbidities with Mortality in COVID-19 Patients: A Systematic Review and Meta-Analysis. Intervirology. 2020 Dec 9:1-12. doi: 10.1159/000512592. Online ahead of print. PMID 33296901
- [Background] Satuan Tugas Penanganan Covid-19. Downloaded from https://covid19.go.id/petasebaran. Accessed 11 October 2021
- [Background] Cirrincione L, Plescia F, Ledda C, Rapisarda V, Martorana D, Moldovan RE, Theodoridou K, Cannizzaro E. COVID-19 Pandemic: Prevention and Protection Measures to Be Adopted at the Workplace. Sustainability 2020; 12: 3603
- [Background] Bloomberg. Downloaded from https://www.bloomberg.com/graphics/covidresilience-ranking/. Accessed 11 October 2021.
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Our world in Data. Downloaded from https://ourworldindata.org/covidvaccinations. Accessed 11 April 2022.
- [Background] CNN. Downloaded from https://edition.cnn.com/2021/04/03/health/uscoronavirus-saturday/index.html. Accessed 11 October 2021.
- [Background] World Health Organization. Downloaded from https://www.who.int/newsroom/feature-stories/detail/vaccine-efficacy-effectiveness-and-protection. Accessed 11 October 2021.
- [Background] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Background] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Background] Reuters. Downloaded from https://www.reuters.com/business/healthcarepharmaceuticals/indonesia-study-finds-chinas-sinovac-covid-19-vaccine-effectivemedical-staff-2021-05-12/. Accessed 11 October 2021
- [Background] Al Kaabi N, Zhang Y, Xia S, Yang Y, Al Qahtani MM, Abdulrazzaq N, Al Nusair M, Hassany M, Jawad JS, Abdalla J, Hussein SE, Al Mazrouei SK, Al Karam M, Li X, Yang X, Wang W, Lai B, Chen W, Huang S, Wang Q, Yang T, Liu Y, Ma R, Hussain ZM, Khan T, Saifuddin Fasihuddin M, You W, Xie Z, Zhao Y, Jiang Z, Zhao G, Zhang Y, Mahmoud S, ElTantawy I, Xiao P, Koshy A, Zaher WA, Wang H, Duan K, Pan A, Yang X. Effect of 2 Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):35-45. doi: 10.1001/jama.2021.8565. PMID 34037666
- [Background] Kyriakidis NC, Lopez-Cortes A, Gonzalez EV, Grimaldos AB, Prado EO. SARS-CoV-2 vaccines strategies: a comprehensive review of phase 3 candidates. NPJ Vaccines. 2021 Feb 22;6(1):28. doi: 10.1038/s41541-021-00292-w. PMID 33619260
- [Background] Mendonca SA, Lorincz R, Boucher P, Curiel DT. Adenoviral vector vaccine platforms in the SARS-CoV-2 pandemic. NPJ Vaccines. 2021 Aug 5;6(1):97. doi: 10.1038/s41541-021-00356-x. PMID 34354082
- [Background] Yadav T, Srivastava N, Mishra G, Dhama K, Kumar S, Puri B, Saxena SK. Recombinant vaccines for COVID-19. Hum Vaccin Immunother. 2020 Dec 1;16(12):2905-2912. doi: 10.1080/21645515.2020.1820808. Epub 2020 Nov 24. PMID 33232211
- [Background] Pollard AJ, Bijker EM. A guide to vaccinology: from basic principles to new developments. Nat Rev Immunol. 2021 Feb;21(2):83-100. doi: 10.1038/s41577-020-00479-7. Epub 2020 Dec 22. PMID 33353987
- [Background] Excler JL, Saville M, Berkley S, Kim JH. Vaccine development for emerging infectious diseases. Nat Med. 2021 Apr;27(4):591-600. doi: 10.1038/s41591-021-01301-0. Epub 2021 Apr 12. PMID 33846611
- [Background] Bhattacharya S, Dasgupta R. Smallpox and polio eradication in India: comparative histories and lessons for contemporary policy. Cien Saude Colet. 2011 Feb;16(2):433-44. doi: 10.1590/s1413-81232011000200007. PMID 21340319
- [Background] CNN Indonesia. Downloaded from https://www.cnnindonesia.com/ekonomi/20210615172504-92-654688/bio-farmayakin-ri-bisa-dapat-400-juta-dosis-vaksin-tahun-ini. Accessed 111 October 2021.
- [Background] Suara.com. Downloaded from https://www.suara.com/bisnis/2020/11/06/151502/ini-6-lembaga-yangkembangkan-vaksin-merah-putih. Accessed 11 October 2021.
- [Background] World Health Organization. Considerations of evaluation of Covid-19 vaccines. Revised. Version of 30 March 2022. Geneva: WHO, 2021.
- [Background] Wang K, Jia Z, Bao L, et al. A subset of Memory B-derived antibody repertoire from 3-dose vaccinees is ultrapotent against diverse and highly transmissible SARS-CoV-2 variants, including Omicron. BioRXiv 2021; doi: https://doi.org/10.1101/2021.12.24.474084;
- [Background] Jara A, Undurraga EA, Gonzalez C, Paredes F, Fontecilla T, Jara G, Pizarro A, Acevedo J, Leo K, Leon F, Sans C, Leighton P, Suarez P, Garcia-Escorza H, Araos R. Effectiveness of an Inactivated SARS-CoV-2 Vaccine in Chile. N Engl J Med. 2021 Sep 2;385(10):875-884. doi: 10.1056/NEJMoa2107715. Epub 2021 Jul 7. PMID 34233097
- [Background] Fonseca MHG, de Souza TFG, de Carvalho Araujo FM, de Andrade LOM. Dynamics of antibody response to CoronaVac vaccine. J Med Virol. 2022 May;94(5):2139-2148. doi: 10.1002/jmv.27604. Epub 2022 Jan 28. PMID 35060174
- [Background] Mascellino MT, Di Timoteo F, De Angelis M, Oliva A. Overview of the Main Anti-SARS-CoV-2 Vaccines: Mechanism of Action, Efficacy and Safety. Infect Drug Resist. 2021 Aug 31;14:3459-3476. doi: 10.2147/IDR.S315727. eCollection 2021. PMID 34511939
- [Background] Prubeta BM. Current State of the First COVID-19 Vaccines. Vaccines (Basel). 2021 Jan 8;9(1):30. doi: 10.3390/vaccines9010030. PMID 33429880
- [Background] Mallapaty S. China's COVID vaccines have been crucial - now immunity is waning. Nature. 2021 Oct;598(7881):398-399. doi: 10.1038/d41586-021-02796-w. No abstract available. PMID 34650240
- [Background] Fadlyana E, Rusmil K, Tarigan R, Rahmadi AR, Prodjosoewojo S, Sofiatin Y, Khrisna CV, Sari RM, Setyaningsih L, Surachman F, Bachtiar NS, Sukandar H, Megantara I, Murad C, Pangesti KNA, Setiawaty V, Sudigdoadi S, Hu Y, Gao Q, Kartasasmita CB. A phase III, observer-blind, randomized, placebo-controlled study of the efficacy, safety, and immunogenicity of SARS-CoV-2 inactivated vaccine in healthy adults aged 18-59 years: An interim analysis in Indonesia. Vaccine. 2021 Oct 22;39(44):6520-6528. doi: 10.1016/j.vaccine.2021.09.052. Epub 2021 Sep 24. PMID 34620531
- [Background] Dinc HO, Saltoglu N, Can G, Balkan II, Budak B, Ozbey D, Caglar B, Karaali R, Mete B, Tuyji Tok Y, Ersoy Y, Ahmet Kuskucu M, Midilli K, Ergin S, Kocazeybek BS. Inactive SARS-CoV-2 vaccine generates high antibody responses in healthcare workers with and without prior infection. Vaccine. 2022 Jan 3;40(1):52-58. doi: 10.1016/j.vaccine.2021.11.051. Epub 2021 Nov 22. PMID 34839992
- [Background] Guzel EC, Celikkol A, Erdal B, Sedef N. Immunogenicity after CoronaVac vaccination. Rev Assoc Med Bras (1992). 2021 Oct;67(10):1403-1408. doi: 10.1590/1806-9282.20210389. PMID 35018966
- [Background] Palacios R, Batista AP, Albuquerque, et al. Efficacy and Safety of a COVID-19 Inactivated Vaccine in Healthcare Professionals in Brazil: The PROFISCOV Study. SSRN 2021; Accessed 3 June 2022. Downoaded at: https://deliverypdf.ssrn.com/delivery.php?ID=840017005024119064102107098125 11906903501500902000007511010309309600701707412300401002803210012605 40480091071111150880671220840550440900110641010140001211230940790260 90054017013015119014069102013003005084113002106123108105096064121107 008029000084020104&EXT=pdf&INDEX=TRUE.
- [Background] Escobar A, Reyes-Lopez FE, Acevedo ML, Alonso-Palomares L, Valiente-Echeverria F, Soto-Rifo R, Portillo H, Gatica J, Flores I, Nova-Lamperti E, Barrera-Avalos C, Bono MR, Vargas L, Simon V, Leiva-Salcedo E, Vial C, Hormazabal J, Cortes LJ, Valdes D, Sandino AM, Imarai M, Acuna-Castillo C. Evaluation of the Immune Response Induced by CoronaVac 28-Day Schedule Vaccination in a Healthy Population Group. Front Immunol. 2022 Jan 31;12:766278. doi: 10.3389/fimmu.2021.766278. eCollection 2021. PMID 35173705
- [Background] Hitchings MDT, Ranzani OT, Torres MSS, de Oliveira SB, Almiron M, Said R, Borg R, Schulz WL, de Oliveira RD, da Silva PV, de Castro DB, Sampaio VS, de Albuquerque BC, Ramos TCA, Fraxe SHH, da Costa CF, Naveca FG, Siqueira AM, de Araujo WN, Andrews JR, Cummings DAT, Ko AI, Croda J. Effectiveness of CoronaVac among healthcare workers in the setting of high SARS-CoV-2 Gamma variant transmission in Manaus, Brazil: A test-negative case-control study. Lancet Reg Health Am. 2021 Sep;1:100025. doi: 10.1016/j.lana.2021.100025. Epub 2021 Jul 25. PMID 34386791
- [Background] De Faria E, Guedes AR, Oliveira MS, et al. Performance of vaccination with CoronaVac in a cohort of healthcare workers (HCW) - preliminary report. MedRXiv 2021; https://doi.org/10.1101/2021.04.12.21255308
- [Background] Ranzani OT, Hitchings MDT, Dorion M, D'Agostini TL, de Paula RC, de Paula OFP, Villela EFM, Torres MSS, de Oliveira SB, Schulz W, Almiron M, Said R, de Oliveira RD, Vieira da Silva P, de Araujo WN, Gorinchteyn JC, Andrews JR, Cummings DAT, Ko AI, Croda J. Effectiveness of the CoronaVac vaccine in older adults during a gamma variant associated epidemic of covid-19 in Brazil: test negative case-control study. BMJ. 2021 Aug 20;374:n2015. doi: 10.1136/bmj.n2015. PMID 34417194
- [Background] Soto JA, Melo-Gozales F, Gutierrez-Vera C, et al. An inactivated SARS-CoV-2 vaccine is safe and induces humoral and cellular immunity against virus variants in healthy children and adolescents in Chile. MedRXiv 2021; https://doi.org/10.1101/2022.02.15.22270973;
- [Background] Schultz BM, Melo-Gonzales, Duarte LF, et al. A booster dose of an inactivated SARS-1 CoV-2 vaccine increases neutralizing antibodies and T cells that recognize Delta and Omicron variants of concern. MedRXiv 2021; https://doi.org/10.1101/2021.11.16.21266350
- [Background] Joko Widodo gets first Sinovac vaccine shot as Indonesia starts mass Covid-19 inoculations. South China Morning Post. Accessed 3 June 2022. Downloaded at: https://www.scmp.com/video/coronavirus/3117548/joko-widodo-gets-first-sinovacvaccine-shot-indonesia-starts-mass-covid
- [Background] Peng Q, Zhou R, Wang Y, Zhao M, Liu N, Li S, Huang H, Yang D, Au KK, Wang H, Man K, Yuen KY, Chen Z. Waning immune responses against SARS-CoV-2 variants of concern among vaccinees in Hong Kong. EBioMedicine. 2022 Mar;77:103904. doi: 10.1016/j.ebiom.2022.103904. Epub 2022 Mar 3. PMID 35248996
- [Background] Chen F, He Y, Shi Y. Parents' and Guardians' Willingness to Vaccinate Their Children against COVID-19: A Systematic Review and Meta-Analysis. Vaccines (Basel). 2022 Jan 24;10(2):179. doi: 10.3390/vaccines10020179. PMID 35214638
- [Background] Walter EB, Talaat KR, Sabharwal C, Gurtman A, Lockhart S, Paulsen GC, Barnett ED, Munoz FM, Maldonado Y, Pahud BA, Domachowske JB, Simoes EAF, Sarwar UN, Kitchin N, Cunliffe L, Rojo P, Kuchar E, Ramet M, Munjal I, Perez JL, Frenck RW Jr, Lagkadinou E, Swanson KA, Ma H, Xu X, Koury K, Mather S, Belanger TJ, Cooper D, Tureci O, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591007 Clinical Trial Group. Evaluation of the BNT162b2 Covid-19 Vaccine in Children 5 to 11 Years of Age. N Engl J Med. 2022 Jan 6;386(1):35-46. doi: 10.1056/NEJMoa2116298. Epub 2021 Nov 9. PMID 34752019
- [Background] Ali K, Berman G, Zhou H, Deng W, Faughnan V, Coronado-Voges M, Ding B, Dooley J, Girard B, Hillebrand W, Pajon R, Miller JM, Leav B, McPhee R. Evaluation of mRNA-1273 SARS-CoV-2 Vaccine in Adolescents. N Engl J Med. 2021 Dec 9;385(24):2241-2251. doi: 10.1056/NEJMoa2109522. Epub 2021 Aug 11. PMID 34379915
- [Background] Han B, Song Y, Li C, Yang W, Ma Q, Jiang Z, Li M, Lian X, Jiao W, Wang L, Shu Q, Wu Z, Zhao Y, Li Q, Gao Q. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine (CoronaVac) in healthy children and adolescents: a double-blind, randomised, controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Dec;21(12):1645-1653. doi: 10.1016/S1473-3099(21)00319-4. Epub 2021 Jun 28. PMID 34197764
- [Background] Chinadaily. Downloaded from: https://www.chinadaily.com.cn/a/202107/20/WS60f60b13a310efa1bd662ea4.html. Accessed at 30 April 2022
- [Background] Pfizer. Dowloaded from: https://www.pfizer.com/news/press-release/press-releasedetail/pfizer-and-biontech-provide-update-rolling-submission. Accessed at 30 April 2022.
- [Background] NBC. Downloaded from: https://www.nbcnews.com/health/health-news/modernaasks-fda-authorize-covid-vaccine-children-6-rcna25816. Accessed at 30 April 2022.